CLINICAL TRIAL: NCT02695602
Title: Prospective Randomized Trial Comparing Microdebrider-Assisted Inferior Turbinoplasty (MAIT) vs Submucous Resection (SMR)
Brief Title: Trial Comparing Microdebrider-Assisted Inferior Turbinoplasty (MAIT) vs Submucous Resection (SMR)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough patients
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-01264
Record Dates: First submitted 2016-02-04; First posted 2016-03-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microdebrider-Assisted Inferior Turbinoplasty (MAIT) (Experimental): Turbinoplasty using microdebrider turbinate blade (2.9mm inferior turbinate blade, Medtronic, 5000 Hz)
  Interventions: Procedure: Microdebrider-Assisted Inferior Turbinoplasty (MAIT)
- Submucous Resection (SMR) (Experimental): Turbinoplasty using non-powered instruments
  Interventions: Procedure: Submucous Resection with non powered instrument

INTERVENTIONS:
Procedure: Microdebrider-Assisted Inferior Turbinoplasty (MAIT)
  Other Names: Medtronic
  Arms: Microdebrider-Assisted Inferior Turbinoplasty (MAIT)
Procedure: Submucous Resection with non powered instrument
  Other Names: Jansen-Middleton or straight through cut
  Arms: Submucous Resection (SMR)

SUMMARY:
This is a prospective, patient blinded, randomized, clinical trial enrolling patients with symptoms and signs of nasal obstruction related to enlarged inferior turbinates. The purpose of this study is to compare two different surgical methods, both of which are already in common use, for the treatment of nasal obstruction in patients with inferior turbinate hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of chronic nasal obstruction with an exam finding of turbinate hypertrophy, with or without septal deviation will be eligible for the study.
* Failed medical treatment
* Have failed medical treatment for at least 1 month, and will be offered surgery
* Patients having Septoplasty at the same time as their turbinate reduction surgery.

Exclusion Criteria:

* Patients who have had previous turbinate reduction surgery will be excluded.
* Patients that have nasal polyps, chronic rhinosinusitis, adenoid hypertrophy, nasal tumors, or any other exam finding that would explain their symptoms of nasal obstruction other than enlarged inferior turbinates with or without septal deviation will be excluded.
* Patients who are diagnosed with purely bony inferior turbinate hypertrophy as discussed below.
* Patients on hormone or anticoagulation therapy and those who have a history of head and neck radiation therapy will be excluded.
* All study candidates will be assessed for external nasal valve collapse via the modified Cottle maneuver, and will be excluded if they exhibit significant external or internal nasal valve collapse as their primary cause of their nasal obstruction.
* All patients will complete the Visual Analog Scale (VAS) on nasal obstruction before and after decongestion at their preoperative visit. Patients that fail to report a score less than 5 after decongestion are likely to have bony rather than soft tissue hypertrophy. In these patients MAIT is unlikely to be an adequate surgical option, and they would derive a greater amount of benefit from SMR. Therefore these patients will be excluded from the study, and offered only SMR.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Nasal Obstruction Symptom Evaluation (NOSE) Score in MAIT vs SMR treated patients | 3 years post-operative
Measure of pain on the Visual Analog Scale | 3 years post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Seth Lieberman, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States